CLINICAL TRIAL: NCT05204498
Title: Efficacy of an Education Plan and Follow-up of Exercise Compliance in Patients With COPD Evaluated Through Knowledge of the Disease With the LINQ Questionnaire and Quality of Life With SGRQ Questionnaire
Brief Title: Efficacy Of An Education Plan And Adherence Follow-Up To The Exercise In Patients With COPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clínica de Occidente S.A (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 0002
Record Dates: First submitted 2019-02-10; First posted 2022-01-24 (Actual); Last update posted 2022-01-24 (Actual); Status verified 2021-11

CONDITIONS: Patient Adherence
Keywords: chronic obstructive pulmonary disease; dyspnea; exercise tolerance; Education
MeSH Terms: conditions — Patient Compliance; Pulmonary Disease, Chronic Obstructive; Dyspnea

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Education plan (Experimental): Education plan and adherence to exercise Educational talk about the importance of exercise as an important strategy to change dyspnea at the start of the study.
  Twice a week, corresponding to the days that do not attend the sessions of pulmonary rehabilitation, calls will be made with a duration of 15 minutes each, in the calls will encourage and guide the practice of physical activity and breathing exercises
  Interventions: Behavioral: Education plan and adherence to exercise
- control (No Intervention): A survey will be conducted at week 8 of monitoring where adherence to exercise is measured during the 8-week study.
  At the end of week 8, patients will be referred to the pulmonary rehabilitation unit in order to evaluate the anthropometric parameters, assess dyspnea with the modified Medical Research Council scale, the hospital anxiety and depression scale, the Saint George respiratory questionnaire, the pulmonary information needs questionnaire and the 6-minute walk test again.

INTERVENTIONS:
Behavioral: Education plan and adherence to exercise — Through phone calls with a motivating sense at any time of the day, twice a week.
  * It will be recorded in an Excel table each time the patient is called.
  * A monthly survey will be applied where the adherence to the exercise during the previous month is measured.
  * These activities will be carried out for 8 weeks. At the end of week 8, patients will be referred to the pulmonary rehabilitation unit to evaluate the anthropometric parameters, assess dyspnea with the modified scale of the Medical Research Council, the hospital anxiety and depression scale, the Saint George respiratory questionnaire , the pulmonary information You need the questionnaire and the 6-minute walk test again.
  Arms: Education plan

SUMMARY:
Chronic obstructive pulmonary disease is one of the main causes of morbidity and mortality worldwide, according to recent publications of the World Health Organization, its main feature is the response to noxious particles of gases, which trigger an inflammatory response with its sequence secondary to the flow of air, the limitation generated by the ventilation reserve mechanism of insufficiency, dyspnea and dysfunction at the muscular level, these limitations generate a high degree of disability worldwide in the different areas of the people who suffer from it, which it affects their basic performance and their interaction with the environment.

The World Health Organization, in a more recent projection, predicted that COPD will increase from its recent classification as the fifth most common cause of mortality to the fourth most common cause by 2030, which would place it behind ischemic cerebrovascular disease, HIV / AIDS and heart disease. More importantly, COPD is a cause that increases chronic disability and is expected to become the fifth most common cause of chronic disability worldwide by 2020.

There is great evidence on the benefit of pulmonary rehabilitation in patients with COPD, which generates changes among which is tolerance to exercise, dyspnea, control of symptoms and improvement in the quality of life related to health. It should be noted that pulmonary rehabilitation not only includes physical training, but also involves the educational component in relation to healthy habits. In this way, patients who have achieved a successful form of a pulmonary rehabilitation program must obtain an improvement in their physical and psychological state, following up on this type of patients, achieving the empowerment of the health process and improving long-term symptoms and healthy lifestyle habits.

Therefore, the objective of this study is to carry out a telephone education and a follow-up plan that emphasizes the importance of physical activity with adequate parameters to be part of the lifestyle of patients and to comply with the activity.

DETAILED DESCRIPTION:
According to the population of the pulmonary rehabilitation center of the private IPS of Cali, it was analyzed by the program coordinator of the Pulmonary Rehabilitation Center.

If you consider that the patient is a candidate to enter the study, you can send an exam to be treated and you can be chosen. If the patient agrees to participate in the study, the knowledge approval process and the application of the clinical route, the basic information of the patient necessary to enter the study is collected.

Once signed, the patient undergoes a physical examination of their clinical and physical condition (Anthropometric parameters, Evaluation of dyspnea with modified scale of the Medical Research Council, Anxiety and Hospital Depression Scale, Saint George Respiratory Questionnaire, needs questionnaire of pulmonary information and 6 minutes walking test).

The walking test that was carried out following the parameters of the American Thoracic Society, in a linear corridor of 30 meters in length, could be used to walk down the corridor for 6 minutes in a row as quickly as possible, vital signs were taken. (blood pressure, heart rate and respiratory rate), oxygen saturation, fatigue in the lower extremities and dyspnea at the beginning and end of the test.

Allocation concealment: the questionnaires, the physical test, the anthropometric parameters were completed and the clinical survey was applied, the information was stored in a closed one and a serial number was assigned according to the order of the exercise. The envelopes were sent to the person responsible for the implementation of the tracking plan that was agreed with the order and the serial number was added to the database.

The randomization of the groups is done in a pre-established template in the following way: simple random sampling with Excel, to list is in the table of the study database and where the variables are collected, the reference number from 1 to 40 according to the number of patients requested to enter the study, apply to a simple randomization formula and a different Excel spreadsheet, up to number 20 (the amount corresponding to the whole follow-up group) B), the numbers that have the The results of this randomization are those assigned to the follow-up group.

In this way, when patients register in the database in the numerical order of the envelope, they are automatically assigned according to the randomization of the group to which the patient belongs (follow-up or control).

Once the patients have been included in the data collection and the variables, the patients belonging to the follow-up group have been submitted to the monitoring monitoring plan, since the activity must be recorded in an Excel table where the control was carried out. and record of it.

The patients attended three times a week, for one hour daily to the pulmonary rehabilitation program to complete a total of 24 sessions, during the sessions the calisthenics were performed, the strengthening of the lower limbs and the strengthening of the upper limbs, the respiratory exercises , continuous exercise for 30 minutes and group and individual educational component during 90 minutes a week, this time of education is in addition to the time of pulmonary rehabilitation.

Once the nursing assistant was responsible for the implementation of the follow-up plan of the process to carry out their activities as follows.

Check the number of patients entering the study, verify the date of admission and the end date, confirm that all patients have cell phones and landlines where they can be located.

She verified that the follow-up charts of each patient were completed, which was done twice a week for a total of 16 follow-ups or 8 weeks of the follow-up plan.

She makes 2 weekly phone calls, performs the days that patients do not attend pulmonary rehabilitation, calls are made with the schedule established in the work template or in the tracking record format.

In each monitoring chart for each patient, the call is recorded, with the recommendations made for patients to perform physical exercise and breathing exercises, the call lasts 15 minutes.

At the end of the 8-week study, Evaluation of Dyspnea with the Scale of the Modified Medical Research Council, The Escalation of Anxiety and Hospital Depression, The Problem of Abortion San Jorge, The Problem of Pulmonary Information Needs and the Walk Test 6 minutes at the Pulmonary Rehabilitation Center.

All the documentation that received the result of the study was guarded by the person in charge of the management of the database and the registry of variables.

The person in charge of the database and the registry of variables is the one who will inform when the study is finished. Subsequently, the information will be organized and the data will be delivered to the methodological advisor to organize, process and analyze the statistical information as a result.

ELIGIBILITY:
Inclusion Criteria:

* Patients clinically stable
* Optimised medical therapy
* Patients who perform pulmonary rehabilitation for the first time
* Postbronchodilator FEV1 < 60% pred and FEV1/forced vital capacity (FVC) < 70% whithout significant reversibility (< 15% change un unutial FEV1)

Exclusion Criteria:

* Clinical evidence of exercise limiting cardiovascular
* Clinical evidence of neuromuscular diseases

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2019-05-10 (Actual); Primary Completion 2019-07-25 (Actual); Study Completion 2019-12-25 (Actual)

PRIMARY OUTCOMES:
Adherence to exercise | Measured at the end of the 8 week monitoring
  practicing physical activity as a principle of self-determination and converting it into a healthy lifestyle or habit and aerobic capacity will be measured by completing 85% of sessions (21 sessions) of pulmonary rehabilitation, including education and telephone follow-up.
knowledge of the disease | Measured at the end of the 8 week monitoring
  Faculty of the human being to understand the aspects related to his illness, the measurement of the needs in education will be carried out through the LINQ Lung Information Needs Questionnaire.
health-related quality of life | Measured at the end of the 8 week monitoring
  A generic concept that reflects the concern for the modification and improvement of the attributes of life, for example, the physical, political, moral, social environment, as well as health and disease.
  It is applied with the Saint George's Questionnaire (SGRQ), this scale goes from 0 to 100 points, high scores indicate that the patient is unwell and low scores the patient is better and a decrease of 4 points after an intervention is considered clinically significant.

CONTACTS AND LOCATIONS:
Overall Officials: Juan Ávila, PT, Principal Investigator — Clínica de Occidente S.A
Locations (1):
- Juan Carlos Avila, Cali, Valle del Cauca Department, Colombia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hill K, Vogiatzis I, Burtin C. The importance of components of pulmonary rehabilitation, other than exercise training, in COPD. Eur Respir Rev. 2013 Sep 1;22(129):405-13. doi: 10.1183/09059180.00002913. PMID 23997066
- [Background] Ávila-Valencia, J. C., Muñoz-Erazo, B. E., Sarria, V., Cordoba, V. B., & Betancourt-Peña, J. (2017). Cambios en el Bode-Bodex de pacientes con EPOC al culminar un programa de rehabilitación pulmonar. Revista colombiana de rehabilitacion, 15(1), 40-47.
- [Background] Vogiatzis I, Nanas S, Roussos C. Interval training as an alternative modality to continuous exercise in patients with COPD. Eur Respir J. 2002 Jul;20(1):12-9. doi: 10.1183/09031936.02.01152001. PMID 12166558
- [Background] Mesquita R, Meijer K, Pitta F, Azcuna H, Goertz YMJ, Essers JMN, Wouters EFM, Spruit MA. Changes in physical activity and sedentary behaviour following pulmonary rehabilitation in patients with COPD. Respir Med. 2017 May;126:122-129. doi: 10.1016/j.rmed.2017.03.029. Epub 2017 Mar 31. PMID 28427543
- [Background] Naseer BA, Al-Shenqiti AM, Ali AH, Al-Jeraisi TM, Gunjan GG, Awaidallah MF. Effect of a short term pulmonary rehabilitation programme on exercise capacity, pulmonary function and health related quality of life in patients with COPD. J Taibah Univ Med Sci. 2017 Aug 23;12(6):471-476. doi: 10.1016/j.jtumed.2017.07.005. eCollection 2017 Dec. PMID 31435281
- [Background] Richards J, Hillsdon M, Thorogood M, Foster C. Face-to-face interventions for promoting physical activity. Cochrane Database Syst Rev. 2013 Sep 30;2013(9):CD010392. doi: 10.1002/14651858.CD010392.pub2. PMID 24085592
- [Background] Hillsdon M, Foster C, Thorogood M. Interventions for promoting physical activity. Cochrane Database Syst Rev. 2005 Jan 25;2005(1):CD003180. doi: 10.1002/14651858.CD003180.pub2. PMID 15674903
- [Background] Aznar S, Webster T. Actividad física y salud en la infancia y la adolescencia: Guía para todas las personas [Internet]. 2006. Available from: http://www.msssi.gob.es/ciudadanos/proteccionSalud/adultos/actiFisica/docs/ActividadFisicaSaludEspanol.pdf
- [Background] Pulmonary rehabilitation: joint ACCP/AACVPR evidence-based guidelines. ACCP/AACVPR Pulmonary Rehabilitation Guidelines Panel. American College of Chest Physicians. American Association of Cardiovascular and Pulmonary Rehabilitation. Chest. 1997 Nov 5;112(5):1363-96. No abstract available. PMID 9367481
- [Background] ATS Committee on Proficiency Standards for Clinical Pulmonary Function Laboratories. ATS statement: guidelines for the six-minute walk test. Am J Respir Crit Care Med. 2002 Jul 1;166(1):111-7. doi: 10.1164/ajrccm.166.1.at1102. No abstract available. PMID 12091180
- [Background] Médicas FDEC, Del R, Hdl C, Carol A, Rojas J. Departamento de Postgrado ANTE EL EJERCICIO FISICO AEROBICO Y ANAEROBICO
- [Background] Gomez LF, Duperly J, Lucumi DI, Gamez R, Venegas AS. [Physical activity levels in adults living in Bogota (Colombia): prevalence and associated factors]. Gac Sanit. 2005 May-Jun;19(3):206-13. doi: 10.1157/13075953. Spanish. PMID 15960953
- [Background] Eden KB, Orleans CT, Mulrow CD, Pender NJ, Teutsch SM. Does counseling by clinicians improve physical activity? A summary of the evidence for the U.S. Preventive Services Task Force. Ann Intern Med. 2002 Aug 6;137(3):208-15. doi: 10.7326/0003-4819-137-3-200208060-00015. PMID 12160371
- [Background] Ilarraza-Lomeli H. [Cardiopulmonary exercise testing]. Arch Cardiol Mex. 2012 Apr-Jun;82(2):160-9. Spanish. PMID 22735657
- [Background] Enright PL, Sherrill DL. Reference equations for the six-minute walk in healthy adults. Am J Respir Crit Care Med. 1998 Nov;158(5 Pt 1):1384-7. doi: 10.1164/ajrccm.158.5.9710086. PMID 9817683